CLINICAL TRIAL: NCT02116764
Title: Analysis of Patients Treated for Chronic Granulomatous Disease Since January 1, 1995
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140091; 14-I-0091
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-19

CONDITIONS: Chronic Granulomatous Disease
Keywords: Rare Diseases; Primary Immune Deficiency Treatment Consortium; Retrospective; Natural History
MeSH Terms: conditions — Granulomatous Disease, Chronic; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cross Sectional: 3 years after Transplant
- No Transplant: These patients were diagnosed with CGD but have not been transplanted
- Prospective: Prior to Transplant Conditioning
- Retrospective: 1 year after Transplant

SUMMARY:
This study is a longitudinal and cross-sectional evaluation of patients with Chronic Granulomatous Disease (CGD) who received or are receiving hematopoietic cell transplantation (HCT) for their disease under a variety of protocols used by participating institutions compared to a control non-HCT group receiving standard care. Investigators at multiple centers caring for patients with CGD in North America and 3 centers in Europe will participate. Patients with CGD will have been treated according to institutional practice and protocols. Investigators will enroll these patients as subjects in this protocol. This study will investigate which patients benefit most from HCT, and what types of transplants are optimal for patients with CGD, in the context of overall outcomes in CGD patients with and without transplant.

DETAILED DESCRIPTION:
This study is a longitudinal and cross-sectional evaluation of patients with Chronic Granulomatous Disease (CGD) who received or are receiving hematopoietic cell transplantation (HCT) for their disease under a variety of protocols used by participating institutions compared to a control non-HCT group receiving standard care. Investigators at multiple centers caring for patients with CGD in North America and 3 centers in Europe will participate. Patients with CGD will have been treated according to institutional practice and protocols. Investigators will enroll these patients as subjects in this protocol. This study will investigate which patients benefit most from HCT, and what types of transplants are optimal for patients with CGD, in the context of overall outcomes in CGD patients with and without transplant.

ELIGIBILITY:
* Both HCT and non-HCT subjects must be over the age of 2 and actively enrolled and receiving treatment under a CGD protocol at NIAID.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with CGD that will be or already Transplanted@@@@@@
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this protocol is to estimate the 1- year, 2-year and 3-year (and longer if possible) overall survival probabilities post-HCT of CGD subjects born on or after 1988 who receive HCTon or after 1995. | 1, 2 or 3 year
  Clinical outcomes (survival, infection, autoimmune disease, chimerism, GVHD)

SECONDARY OUTCOMES:
To compare overall survival from birth between patients born on or after 1988 who receive HCT on or after 1995 vs. those born on or after 1988 who receive conventional therapy, after adjusting for differences in year of birth and oxidase acti... | 3 years post Transplant or Non Transplant
  Clinical outcomes (survival, infection, autoimmune disease, chimerism, GVHD)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kuhns DB, Alvord WG, Heller T, Feld JJ, Pike KM, Marciano BE, Uzel G, DeRavin SS, Priel DA, Soule BP, Zarember KA, Malech HL, Holland SM, Gallin JI. Residual NADPH oxidase and survival in chronic granulomatous disease. N Engl J Med. 2010 Dec 30;363(27):2600-10. doi: 10.1056/NEJMoa1007097. PMID 21190454
- [Background] Kobayashi S, Murayama S, Takanashi S, Takahashi K, Miyatsuka S, Fujita T, Ichinohe S, Koike Y, Kohagizawa T, Mori H, Deguchi Y, Higuchi K, Wakasugi H, Sato T, Wada Y, Nagata M, Okabe N, Tatsuzawa O. Clinical features and prognoses of 23 patients with chronic granulomatous disease followed for 21 years by a single hospital in Japan. Eur J Pediatr. 2008 Dec;167(12):1389-94. doi: 10.1007/s00431-008-0680-7. Epub 2008 Mar 12. PMID 18335239
- [Background] Gallin JI, Alling DW, Malech HL, Wesley R, Koziol D, Marciano B, Eisenstein EM, Turner ML, DeCarlo ES, Starling JM, Holland SM. Itraconazole to prevent fungal infections in chronic granulomatous disease. N Engl J Med. 2003 Jun 12;348(24):2416-22. doi: 10.1056/NEJMoa021931. PMID 12802027
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-I-0091.html